CLINICAL TRIAL: NCT03532516
Title: Compassionate Use Program With Brivaracetam for the Treatment of Patients With Epilepsy
Status: Available | Type: Expanded Access
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: N01317
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Brivaracetam — Patients will start on the individual Brivaracetam (BRV) dose that they had reached at the completion of the previous study. The BRV dose can be adjusted based on the individual patient's seizure control and tolerability; however, the BRV dose may not exceed 200 mg/day in divided (preferably symmetrical) morning and evening doses, taken with or without food.
  Up- and down-titration steps should be performed in steps of maximum 50 mg/day on a weekly basis. The full down-titration should include a 1-week step at 20 mg/day.
  Other Names: Briviact

SUMMARY:
This Compassionate Use Program (CUP) is setup to provide study patients with continuous access to Brivaracetam (BRV) for the time period between closures of the long-term follow up studies N01125, N01199, N01372, N01379, and N01315 and when BRV is commercially available.

ELIGIBILITY:
Inclusion Criteria:

* Patients with epilepsy who are participating in Brivaracetam (BRV) studies N01125, N01199, N01372, N01379 or N01315
* Patients for whom the treating physician believes there is a continued benefit from the long-term administration of BRV and other anti-epileptic therapies might not be suitable for the patient
* Female patients without childbearing potential are eligible
* Female patients with childbearing potential are eligible if they use a medically accepted contraceptive method for the duration of the Compassionate Use Program (CUP) participation. The patient must understand the consequences and potential risks of inadequately protected sexual activity, be educated about and understand the proper use of contraceptive methods, and inform the treating physician of any potential change in status
* Patient is considered reliable and capable of adhering to medication intake.
* Patient is informed of the details of this CUP, is given ample time and opportunity to ask questions and consider his/her participation in this CUP, and the patient or the legally authorized representative (LAR) has provided verbal consent to participate, and, if required under local regulations, has given written informed consent

Exclusion Criteria:

* Severe medical, neurological and psychiatric disorders, including current suicidal ideation or behavior, or laboratory values which may have an impact on the safety of the patient, as determined by the treating physician
* Poor compliance with medication intake in the previous BRV study
* Participation in any clinical study of another investigation drug or device during the CUP
* Pregnant or lactating woman

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)